CLINICAL TRIAL: NCT07112911
Title: Restoring Functional Capacity of the Upper Extremity Using Combined Neuromuscular Electrical Stimulation Robot and Trans-Spinal Electrical Stimulation in Individuals With Chronic Stroke
Brief Title: Effects of Combined Neuromuscular Electrical Stimulation Robot and Trans-Spinal Electrical Stimulation in Poststroke Rehabilitation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Xiaoling Hu, Director of Research Postgraduate Studies and Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSEARS20250520004
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Electric Stimulation; Occupational Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tsES-ENMS rehabilitation (Experimental): The stroke participants will receive trans-spinal electrical stimulation (tsES), peripheral activation via neuromuscular electrical stimulation (NMES), and task-specific upper limb robotic training. A mobile hybrid neuromuscular electrical stimulation (NMES)-robot, i.e., exoneuromusculoskeleton (ENMS) was adopted in the experiment.
  Interventions: Device: Electrical Stimulation; Rehabilitation Robot
- tsES-OT rehabilitation (Active Comparator): The stroke participants will receive a task-oriented occupational therapy(OT), along with trans-spinal electrical stimulation (tsES) rehabilitation.
  Interventions: Behavioral: Occupational Therapy with Electrical Stimulation
- sham tsES-OT rehabilitation (Sham Comparator): The stroke participants will receive a task-oriented occupational therapy, along with sham trans-spinal electrical stimulation (tsES) rehabilitation.
  Interventions: Behavioral: occupational therapy with sham electrical stimulation

INTERVENTIONS:
Device: Electrical Stimulation; Rehabilitation Robot — The recruited subjects will receive 20 sessions of robot-assisted upper limb training combined with central-to-peripheral electrical stimulation, delivered at a frequency of 3 to 5 sessions per week, which will be completed within 4 to 7 consecutive weeks. Each rehabilitation session will begin with a 10-minute preparation phase, followed by 20 minutes of NMES and tsES-assisted robotic training. After a 10-minute break, the session will continue with an additional 20 minutes of robotic-assisted training combined with NMES alone, with tsES turned off during this phase. During the training, patients will perform repeated wrist and finger flexion-extension tasks. The training protocol is designed to activate wrist extension voluntarily (exceeding 10% of their initial MVC), which then triggers NMES and inflation of the robotic hand to assist finger opening.
  Arms: tsES-ENMS rehabilitation
Behavioral: Occupational Therapy with Electrical Stimulation — The recruited subjects will receive 20 sessions of task-oriented occupational therapy(OT) combined with trans-spinal electrical stimulation(tsES), delivered at a frequency of 3 to 5 sessions per week, which will be completed within 4 to 7 consecutive weeks. Each rehabilitation session will begin with a 10-minute preparation phase, followed by 20 minutes of OT training with tsES. After a 10-minute break, the session will continue with an additional 20 minutes of COT alone, with tsES turned off during this phase. During the OT training, the stroke participants will perform functional daily living tasks, including cylindrical grasp, disc grasp, and tip pinch.
  Arms: tsES-OT rehabilitation
Behavioral: occupational therapy with sham electrical stimulation — The recruited subjects will receive 20 sessions of task-oriented occupational therapy(OT) combined with sham trans-spinal electrical stimulation(tsES), delivered at a frequency of 3 to 5 sessions per week, which will be completed within 4 to 7 consecutive weeks. Each rehabilitation session will begin with a 10-minute preparation phase, followed by 20 minutes of OT training with 0mA-intensity tsES. After a 10-minute break, the session will continue with an additional 20 minutes of COT alone, with tsES turned off during this phase. During the training, the stroke participants will repeatedly practice functional daily living tasks, including cylindrical grasp, disc grasp, and tip pinch.
  Arms: sham tsES-OT rehabilitation

SUMMARY:
The purpose of this study is to investigate the clinical efficacy and neurological progress of combined training using trans-spinal electrical stimulation (tsES) and neuromuscular electrical stimulation (NMES)-driven robotics on upper limb rehabilitation after stroke

DETAILED DESCRIPTION:
This study aims to explore whether a multimodal intervention that combines central neuromodulation through trans-spinal electrical stimulation (tsES), peripheral activation via neuromuscular electrical stimulation (NMES), and task-specific robotic training can enhance upper limb recovery.

Specific objectives:

1. To evaluate the clinical efficacy of combining tsES and NMES robotic training for enhancing upper limb motor function in post-stroke patients.
2. To quantify the neurological progress of the tsES and NMES robot combined interventions in the rehabilitation process using electrophysiological tracers (electroencephalogram, electromyogram) and kinesiological recorder (Inertial Measurement Unit)
3. To investigate the central-to-peripheral neuroplasticity by corticomuscular coherence evaluation in poststroke rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* Subjects in the chronic stage (start from 6 months after the onset of stroke) with a pure unilateral motor paresis after a stroke (ischemic or hemorrhagic);
* Sufficient cognition to follow simple instructions as well as understand the content and purpose of the experiment (Mini-Mental State Examination (MMSE) score>23);
* Be able to sit up for 60 minutes (with or without assistance);
* Muscle strength graded from 1 to 3 in biceps brachii, triceps brachii, extensor carpi radialis, flexor carpi radialis, and abductor pollicis brevis in the affected side.
* The voluntary electromyographic signals of the wrist extensor and wrist flexor muscle groups can be detected.

Exclusion Criteria:

* Patients with secondary stroke;
* Severe dysphasia (either expressive or comprehensive) with inadequate communication;
* Any additional medical or psychological condition affecting their ability to comply with the study protocol;
* History of other neurological disease, psychiatric disorder, including alcoholism and substance abuse;
* currently pregnant;
* epilepsy;
* pacemaker implantation or deep brain stimulation;
* involved in drug studies, other clinical trials, or concurrent medication/occupational/physical treatments on the upper limb;
* skin disease at the area of the electrodes;
* High hypertension and cannot maintain normal blood pressure despite daily intake of antihypertensive medication.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment Scale after training | Within 1 week before the start of training Within 1 week after the completion of training 3 months after the completion of training
  The Fugl-Meyer Assessment (FMA) Scale for the upper limb measures voluntary motor function in the shoulder, wrist, and hand. The total score ranges from 0 to 66, with higher scores indicating better motor function. The scale can be further divided into two subscores: shoulder/elbow (0-42) and wrist/hand (0-24).

SECONDARY OUTCOMES:
Change in Modified Ashworth Scale(MAS), Action Research Arm Test (ARAT), Wolf Motor Function Test (WMFT) after training | Within 1 week before the start of training Within 1 week after the completion of training 3 months after the completion of training
  The Modified Ashworth Scale (MAS) assesses muscle spasticity by measuring resistance during passive joint movement, particularly in the flexor muscles. The MAS consists of six levels, ranging from 0 to 4 (with an additional grade of 1+), where higher scores indicate increased resistance and greater muscle spasticity.
  The Action Research Arm Test (ARAT) evaluates upper limb motor function by measuring the ability to perform specific tasks related to grasp, grip, pinch, and gross movement. It consists of 19 items, each scored from 0 to 3, with a total score ranging from 0 to 57. Higher scores represent better upper limb functional performance.
  The Wolf Motor Function Test (WMFT) assesses upper extremity motor ability through a series of timed and functional tasks. It includes 15 function-based items and 2 strength-based items. Each task is timed and rated on a 6-point functional ability scale, where higher scores and faster completion times reflect better motor performance.
Change in Cortico-Muscular Coherence (CMC) after training | Within 1 week before the start of training Within 1 week after the completion of training 3 months after the completion of training
  Cortico-Muscular Coherence (CMC) is calculated using simultaneous EEG and EMG recordings to assess the functional connectivity between the motor cortex and the target muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoling HU, Principal Investigator — The Hong Kong Polyterchnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided